CLINICAL TRIAL: NCT00526006
Title: PPI-Rebound-Trial. A Study of the Clinical Relevance of the Acid Rebound Phenomena
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-00673-145
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2007-09-06 (Estimated); Status verified 2007-08

CONDITIONS: Healthy
Keywords: Clinical significance of the acid rebound phenomenon after withdrawal of treatment with a PPI
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: esomeprazole — 40 mg od for 8 wks

SUMMARY:
The acid secretion in the stomach seems to increase after withdrawal of min. 8 wks of treatment with a PPI (protonpump inhibitor) It is unknown if this acid rebound phenomenon is of clinical significance. In a doubleblinded and placebocontrolled study healthy volunteers are randomized to treatment with placebo or PPI + placebo. Gastrointestinal symptoms are scored once a week and.

ELIGIBILITY:
Inclusion Criteria:

* 18 years +

Exclusion Criteria:

* Dyspepsia, heartburn og acid regurgitation within the preceeding 4 weeks
* Previous treatment with PPI og H2RA
* Previous contact to doctor or hospital because of dyspepsia or reflux
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-09; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Symptom scores in the reflux part of the GSRS after withdrawal of active treatment in the actively treated group versus the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Christina Reimer, MD, Principal Investigator — University Hospital Køge
Locations (1):
- University Hospital Køgw, Køge, Denmark